CLINICAL TRIAL: NCT05819658
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Design, Prospective, Phase IIa Exploratory Clinical Trial to Evaluate the Efficacy and Safety of SC Administration of GV1001 0.56 or 1.12 mg/Day in Patients With PSP
Brief Title: GV1001 Subcutaneous(SC) for the Treatment of Progressive Supranuclear Palsy (PSP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GemVax & Kael (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GV1001-PSP-CL2-011
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Progressive Supranuclear Palsy
Keywords: Progressive Supranuclear Palsy; GV1001
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo SC injection will be administered once weekly for 4 weeks then every 2 weeks through Week 24 for double blind phase.
  Interventions: Drug: GV1001 Placebo
- GV1001 0.56 mg (Experimental): GV1001 0.56 mg SC injection will be administered once weekly for 4 weeks then every 2 weeks through Week 24 for double blind phase.
  Interventions: Drug: GV1001 0.56mg
- GV1001 1.12 mg (Experimental): GV1001 1.12 mg SC injection administered once weekly for 4 weeks then every 2 weeks through Week 24 for double blind phase.
  Interventions: Drug: GV1001 1.12mg

INTERVENTIONS:
Drug: GV1001 Placebo — 0.9% normal saline
  Other Names: Normal saline
  Arms: Placebo
Drug: GV1001 0.56mg — Lyophilized peptide from hTERT
  Other Names: Tertomotide 0.84mg
  Arms: GV1001 0.56 mg
Drug: GV1001 1.12mg — Lyophilized peptide from hTERT
  Other Names: Tertomotide 1.68mg
  Arms: GV1001 1.12 mg

SUMMARY:
The study will be conducted by the Sponsor to evaluate the efficacy and safety of GV1001 (0.56 mg and 1.12 mg) administered subcutaneously as a treatment for Progressive Supranuclear Palsy, (PSP). In 75 patients diagnosed with PSPR Richardson(PSP-RS) or PSP-Parkinsonism (PSP-P) at five hospitals in Korea, subcutaneous administration of GV1001 0.56 or 1.12 mg/day will be conducted with multicenter, randomized, double-blind, placebo-controlled, parallel design, prospective phase 2a.

DETAILED DESCRIPTION:
This is a 24-week, multicenter, randomized, double-blind, placebo-controlled, parallel design, prospective, Phase 2a exploratory clinical study. If the subject and/or the subject's representative provide a written consent to participate in this clinical study, the required examinations and tests will be performed at the screening visit, and the screening period will run for 4 weeks or shorter. Subjects who are ultimately determined as eligible by the inclusion/exclusion criteria after screening will be randomized at a 1:1:1 ratio to Study Group 1 (GV1001 0.56 mg/day), Study Group 2 (GV1001 1.12 mg/day), or the placebo group depending on the study site in which they are enrolled. Depending on the randomization results, subjects will be administered the investigational product (study drug or placebo) once weekly for the first 4 weeks (1 month), and then administered 10 times at 2-week intervals for 20 weeks (5 months) for a total of 14 doses over 24 weeks (6 months). All subjects will visit the institution according to the planned clinical study schedule to receive the investigational product and to be evaluated for efficacy and safety. To ensure the objectivity and accuracy of the study results, the individuals evaluating efficacy will be limited to neurologists who have been sufficiently educated and trained, and the collection of efficacy and safety evaluation data and biomarkers will be performed in a consistent order at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥41 years to ≤ 85 years.
* Clinical diagnosis of probable progressive supranuclear palsy (PSP).
* Patient is on a stable therapy for a neurological drug for at least 1 month prior to screening visit.
* Patients who are able to walk 3 meters or more independently or with assistive devices.
* Score 15 points ≥ on the Korean Mini-Mental Status Exam (K-MMSE) at the screening visit.
* Have reliable caregiver to accompany participant to all study visits.
* Patients and/or their representatives who have voluntarily provided a written consent for participation in this clinical study.

Exclusion Criteria:

* Patients who have Presence of structural lesions or Suspected concurrent onset of central nervous system diseases based on the CT/MRI scan results and neurological examinations performed within 12 months of screening or at screening.
* Patients with a history of known or suspected seizures.
* Patients with a recent unexplained loss of consciousness within 3 months prior to screening or a history of significant head trauma with loss of consciousness.
* Patients with acute or unstable cardiovascular disease, uncontrolled hypertension, uncontrolled diabetes, or any other medical condition that can interfere with completing the clinical study.
* Patients with hypersensitivity reactions to the ingredients of the investigational product.
* Patients with a history of cancer within 5 years prior to screening.
* Patients with abnormal renal function.
* Patients with severe liver function abnormalities.
* Patients weighing ≤35 kg.
* Among the female subjects who does not agree to use proper contraception.
* Pregnant or breastfeeding women.
* Patients who participated in another clinical study within 4 weeks prior to screening and were administered investigational products or were applied investigational medical devices.
* Patients who were administered the study drug (GV1001) of this clinical study within 12 months prior to screening.
* Patients who participated in a clinical study for progressive supranuclear palsy within 6 months prior to screening.
* Other patients judged by the investigator as ineligible to participate in this clinical study.

Ages: 41 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Jae Kim, Study Chair — GemVax & Kael
Locations (5):
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kyung Hee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Started | 25 | 25 | 28
Completed | 22 | 20 | 25
Not Completed | 3 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg | Total
Number analyzed (Participants) | 25 | 25 | 28 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 6 | 26
  Male | 14 | 16 | 22 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 25 | 25 | 28 | 78
PSP type [Count of Participants; unit: Participants] — PSP-RS type: patients with clearly identified supranuclear ophthalmoplegia (SOP) according to the judgment of the investigator.
  PSP-p type: patients identified as having shown little or no response to previous administration of levodopa according to the judgment of the investigator.
  Participants
    PSP-Richardson type | 18 | 16 | 21 | 55
    PSP Parkinsonian type | 7 | 9 | 7 | 23
Age, Categorical [Count of Participants; unit: Participants] — Participants aged 41 to 85 years old
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 6 | 7 | 3 | 16
    >=65 years | 19 | 18 | 25 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change From the Baseline in the Total Score of PSP-rating Scale
Description: Change from the baseline in the total score of PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 24 weeks (6 months) of investigational product administration. The possible total scores range from 0 to 100 with a higher score indicating severely impaired cognitive function.
Time Frame: 24 weeks(6 months)
Population: Participants who completed 24 weeks (6 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 20 | 25
scores on a scale | 4.10 (1.69) | 2.14 (1.78) | 6.46 (1.64)

2. Secondary Outcome: Change From the Baseline in the Total Score of PSP-rating Scale
Description: Change from the baseline in the total score of PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 12 weeks (3 months) of investigational product administration. The possible total scores range from 0 to 100 with a higher score indicating severely impaired cognitive function.
Time Frame: 12 Weeks(3 months)
Population: Participants who completed 12 weeks (3 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 22 | 26
scores on a scale | 1.42 (1.60) | -0.47 (1.65) | 2.75 (1.55)

3. Secondary Outcome: Change From the Baseline in the Montreal Cognitive Assessment - Korea (MoCAK)
Description: Change from the baseline in the Montreal Cognitive Assessment - Korea (MoCAK) after 12 weeks (3 months) of investigational product administration. The possible total scores range from 0 to 30 with a higher score indicating greater cognitive function.
Time Frame: 12 weeks (3 Months)
Population: Participants who completed 12 weeks (3 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 22 | 26
scores on a scale | 0.25 (0.61) | 0.93 (0.64) | 0.26 (0.60)

4. Secondary Outcome: Change From the Baseline in the Montreal Cognitive Assessment - Korea (MoCAK)
Description: Change from the baseline in the Montreal Cognitive Assessment - Korea (MoCAK) after 24 weeks (6 months) of investigational product administration. The possible total scores range from 0 to 30 with a higher score indicating greater cognitive function.
Time Frame: 24 weeks(6 months)
Population: Participants who completed 24 weeks (6 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 20 | 25
scores on a scale | 0.29 (0.73) | 0.35 (0.78) | -1.46 (0.71)

5. Secondary Outcome: Change From the Baseline in the Korean Frontal Assessment Battery (K-FAB)
Description: Change from the baseline in the Korean Frontal Assessment Battery (K-FAB) after 12 weeks (3 months) of investigational product administration. The possible total scores range from 0 to 18 with a higher score indicating greater cognitive function.
Time Frame: 12 weeks(3 months)
Population: Participants who completed 12 weeks (3 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 22 | 26
scores on a scale | -0.29 (0.51) | -1.06 (0.53) | -1.42 (0.49)

6. Secondary Outcome: Change From the Baseline in the Korean Frontal Assessment Battery (K-FAB)
Description: Change from the baseline in the Korean Frontal Assessment Battery (K-FAB) after 24 weeks (6 months) of investigational product administration. The possible total scores range from 0 to 18 with a higher score indicating greater cognitive function.
Time Frame: 24 weeks(6 months)
Population: Participants who completed 24 weeks (6 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 20 | 25
scores on a scale | -0.20 (0.55) | -0.89 (0.59) | -1.42 (0.54)

7. Secondary Outcome: Change From the Baseline in the England & Schwab Activity of Daily Living (ES ADL) Scale
Description: Change from the baseline in the England & Schwab Activity of Daily Living (ES ADL) scale after 12 weeks (3 months) of investigational product administration. The possible total scores range from 0 (complete dependence) to 100% (complete independence) based on the level of independence.
Time Frame: 12 weeks(3 months)
Population: Participants who completed 12 weeks (3 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 22 | 26
scores on a scale | -2.18 (2.92) | -2.70 (3.02) | -7.12 (2.85)

8. Secondary Outcome: Change From the Baseline in the England & Schwab Activity of Daily Living (ES ADL) Scale
Description: Change from the baseline in the England & Schwab Activity of Daily Living (ES ADL) scale after 24 weeks (6 months) of investigational product administration. The possible total scores range from 0 (complete dependence) to 100% (complete independence) based on the level of independence.
Time Frame: 24 weeks(6 months)
Population: Participants who completed 24 weeks (6 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 20 | 25
scores on a scale | -9.45 (3.05) | -8.35 (3.23) | -17.12 (2.99)

9. Secondary Outcome: Change From the Baseline in the Score of Each Domain of the PSP-rating Scale (History)
Description: Change from the baseline in the score of [History] domain of the PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 12 weeks (3 months) of investigational product administration. The possible total scores range from 0 to 24 with a higher score indicating severely impaired cognitive function.
Time Frame: 12 weeks(3 months)
Population: Participants who completed 12 weeks (3 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 22 | 26
scores on a scale | -0.26 (0.56) | -0.17 (0.59) | 0.41 (0.55)

10. Secondary Outcome: Change From the Baseline in the Score of Each Domain of the PSP-rating Scale (History)
Description: Change from the baseline in the score of [History] domain of the PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 24 weeks (6 months) of investigational product administration. The possible total scores range from 0 to 24 with a higher score indicating severely impaired cognitive function.
Time Frame: 24 weeks(6 months)
Population: Participants who completed 24 weeks (6 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 20 | 25
scores on a scale | 0.42 (0.66) | 0.90 (0.70) | 1.36 (0.64)

11. Secondary Outcome: Change From the Baseline in the Score of Each Domain of the PSP-rating Scale (Mentation)
Description: Change from the baseline in the score of [Mentation] domain of the PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 12 weeks (3 months) of investigational product administration. The possible total scores range from 0 to 16 with a higher score indicating severely impaired cognitive function.
Time Frame: 12 weeks(3 months)
Population: Participants who completed 12 weeks (3 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 22 | 26
scores on a scale | 0.31 (0.41) | -0.01 (0.41) | 0.23 (0.39)

12. Secondary Outcome: Change From the Baseline in the Score of Each Domain of the PSP-rating Scale (Mentation)
Description: Change from the baseline in the score of [Mentation] domain of the PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 24 weeks (6 months) of investigational product administration. The possible total scores range from 0 to 16 with a higher score indicating severely impaired cognitive function.
Time Frame: 24 weeks(6 months)
Population: Participants who completed 24 weeks (6 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 20 | 25
scores on a scale | 0.26 (0.41) | -0.07 (0.43) | 0.66 (0.40)

13. Secondary Outcome: Change From the Baseline in the Score of Each Domain of the PSP-rating Scale (Bulbar)
Description: Change from the baseline in the score of [Bulbar] domain of the PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 12 weeks (3 months) of investigational product administration. The possible total scores range from 0 to 8 with a higher score indicating severely impaired cognitive function.
Time Frame: 12 weeks(3 months)
Population: Participants who completed 12 weeks (3 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 22 | 26
scores on a scale | 0.35 (0.24) | 0.11 (0.25) | -0.08 (0.24)

14. Secondary Outcome: Change From the Baseline in the Score of Each Domain of the PSP-rating Scale (Bulbar)
Description: Change from the baseline in the score of [Bulbar] domain of the PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 24 weeks (6 months) of investigational product administration. The possible total scores range from 0 to 8 with a higher score indicating severely impaired cognitive function.
Time Frame: 24 weeks(6 months)
Population: Participants who completed 24 weeks (6 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 20 | 25
scores on a scale | 0.49 (0.26) | 0.04 (0.28) | 0.68 (0.26)

15. Secondary Outcome: Change From the Baseline in the Score of Each Domain of the PSP-rating Scale (Ocular Motor)
Description: Change from the baseline in the score of [Ocular Motor] domain of the PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 12 weeks (3 months) of investigational product administration. The possible total scores range from 0 to 16 with a higher score indicating severely impaired cognitive function.
Time Frame: 12 weeks(3 months)
Population: Participants who completed 12 weeks (3 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 22 | 26
scores on a scale | -0.05 (0.48) | 0.08 (0.49) | 0.86 (0.46)

16. Secondary Outcome: Change From the Baseline in the Score of Each Domain of the PSP-rating Scale (Ocular Motor)
Description: Change from the baseline in the score of [Ocular Motor] domain of the PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 24 weeks (6 months) of investigational product administration. The possible total scores range from 0 to 16 with a higher score indicating severely impaired cognitive function.
Time Frame: 24 weeks(6 months)
Population: Participants who completed 24 weeks (6 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 20 | 25
scores on a scale | 1.36 (0.44) | 0.25 (0.46) | 1.30 (0.43)

17. Secondary Outcome: Change From the Baseline in the Score of Each Domain of the PSP-rating Scale (Limb Motor)
Description: Change from the baseline in the score of [Limb Motor] domain of the PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 12 weeks (3 months) of investigational product administration. The possible total scores range from 0 to 16 with a higher score indicating severely impaired cognitive function.
Time Frame: 12 weeks(3 months)
Population: Participants who completed 12 weeks (3 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 22 | 26
scores on a scale | 0.27 (0.36) | -0.26 (0.38) | 0.02 (0.36)

18. Secondary Outcome: Change From the Baseline in the Score of Each Domain of the PSP-rating Scale (Limb Motor)
Description: Change from the baseline in the score of [Limb Motor] domain of the PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 24 weeks (6 months) of investigational product administration. The possible total scores range from 0 to 16 with a higher score indicating severely impaired cognitive function.
Time Frame: 24 weeks(6 months)
Population: Participants who completed 24 weeks (6 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 20 | 25
scores on a scale | 0.45 (0.52) | -0.07 (0.55) | 0.51 (0.50)

19. Secondary Outcome: Change From the Baseline in the Score of Each Domain of the PSP-rating Scale (Midline/Gait)
Description: Change from the baseline in the score of [Midline/Gait] domain of the PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 12 weeks (3 months) of investigational product administration. The possible total scores range from 0 to 20 with a higher score indicating severely impaired cognitive function.
Time Frame: 12 weeks(3 months)
Population: Participants who completed 12 weeks (3 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 22 | 26
scores on a scale | 0.26 (0.47) | -0.08 (0.49) | 1.19 (0.46)

20. Secondary Outcome: Change From the Baseline in the Score of Each Domain of the PSP-rating Scale (Midline/Gait)
Description: Change from the baseline in the score of [Midline/Gait] domain of the PSP-rating scale(Progressive Supranuclear Palsy Rating Scale) after 24 weeks (6 months) of investigational product administration. The possible total scores range from 0 to 20 with a higher score indicating severely impaired cognitive function.
Time Frame: 24 weeks(6 months)
Population: Participants who completed 24 weeks (6 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 20 | 25
scores on a scale | 0.58 (0.56) | 1.28 (0.59) | 1.79 (0.54)

21. Secondary Outcome: Change From the Baseline in the Score of Each Item of the PSP-rating Scale(Item 12_Dysarthria)
Description: Change from the baseline in the score of each item [Item 12_Dysarthria] of the PSP-rating scale after 12 weeks (3 months) of investigational product administration. Only the analysis result for Item no.12 out of a total of 28 items is described. The possible total scores range from 0 to 4 with a higher score indicating severely impaired cognitive function.
Time Frame: 12 weeks(3 months)
Population: Participants who completed 12 weeks (3 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 22 | 26
scores on a scale | 0.21 (0.15) | 0.13 (0.15) | 0.06 (0.14)

22. Secondary Outcome: Change From the Baseline in the Score of Each Item of the PSP-rating Scale(Item 12_Dysarthria)
Description: Change from the baseline in the score of each item [Item 12_Dysarthria] of the PSP-rating scale after 24 weeks (6 months) of investigational product administration. Only the analysis result for Item no.12 out of a total of 28 items is described. The possible total scores range from 0 to 4 with a higher score indicating severely impaired cognitive function.
Time Frame: 24 weeks(6 months)
Population: Participants who completed 24 weeks (6 months) were included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
Number analyzed (Participants) | 22 | 20 | 25
scores on a scale | 0.44 (0.14) | 0.01 (0.15) | 0.44 (0.14)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 28 weeks
Description: Participants who were not treated were excluded.(0.56mg/day group: 1. Placebo group: 1)
Arm/Group | Placebo | GV1001 0.56 mg | GV1001 1.12 mg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/28
Serious Adverse Events (participants affected / at risk) | 3/24 | 2/24 | 5/28
Other Adverse Events (participants affected / at risk) | 15/24 | 12/24 | 9/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | GV1001 0.56 mg (N=24) | GV1001 1.12 mg (N=28)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Infective spondylitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tuberculous pleurisy (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | GV1001 0.56 mg (N=24) | GV1001 1.12 mg (N=28)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 2 (11) | 1 (4) | 3 (9)
Chest pain (General disorders) | 3 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT05819658/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT05819658/SAP_001.pdf